CLINICAL TRIAL: NCT01004822
Title: A Phase 1, Multicenter, Open-label, Dose-escalation, Safety, Pharmacokinetic, And Pharmacodynamic Study Of Cvx-241, A Selective Angiopoietin-2 And Vascular Endothelial Growth Factor Binding, Anti-angiogenic Covx-body, In Patients With Advanced Solid Tumors
Brief Title: A Safety, Tolerability, And Pharmacokinetic Trial With CVX-241 In Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1561001; CVX-241-101 (Other: Alias Study Number)
Record Dates: First submitted 2009-10-28; First posted 2009-10-30 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Advanced Solid Tumors
Keywords: Treatment Non-Randomized Single Group Assignment Safety Study Neoplasms Carcinoma Cancer Malignancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Drug (Experimental): Weekly infusions of CVX-241 at specified doses
  Interventions: Drug: CVX-241

INTERVENTIONS:
Drug: CVX-241 — 0.3 mg/kg infusions of CVX-241 on Days 1, 8, 15, and 22 of each 28 day cycle. Weekly infusions administered until progression or unacceptable toxicity develops.
  Other Names: PF-05057459
Drug: CVX-241 — 1 mg/kg infusions of CVX-241 on Days 1, 8, 15, and 22 of each 28 day cycle. Weekly infusions administered until progression or unacceptable toxicity develops.
  Other Names: PF-05057459
Drug: CVX-241 — 3 mg/kg infusions of CVX-241 on Days 1, 8, 15, and 22 of each 28 day cycle. Weekly infusions administered until progression or unacceptable toxicity develops.
  Other Names: PF-05057459
Drug: CVX-241 — 6 mg/kg infusions of CVX-241 on Days 1, 8, 15, and 22 of each 28 day cycle. Weekly infusions administered until progression or unacceptable toxicity develops.
  Other Names: PF-05057459
Drug: CVX-241 — 12 mg/kg infusions of CVX-241 on Days 1, 8, 15, and 22 of each 28 day cycle. Weekly infusions administered until progression or unacceptable toxicity develops.
  Other Names: PF-05057459
Drug: CVX-241 — 15 mg/kg infusions of CVX-241 on Days 1, 8, 15, and 22 of each 28 day cycle. Weekly infusions administered until progression or unacceptable toxicity develops.
  Other Names: PF-05057459
Drug: CVX-241 — 18 mg/kg infusions of CVX-241 on Days 1, 8, 15, and 22 of each 28 day cycle. Weekly infusions administered until progression or unacceptable toxicity develops.
  Other Names: PF-05057459
Drug: CVX-241 — 25 mg/kg infusions of CVX-241 on Days 1, 8, 15, and 22 of each 28 day cycle. Weekly infusions administered until progression or unacceptable toxicity develops.
  Other Names: PF-05057459

SUMMARY:
The purpose of this study is to determine if CVX-241 (PF-05057459) is safe and tolerable when given as weekly infusions to adult patients with advanced solid tumors.

DETAILED DESCRIPTION:
The study was prematurely discontinued on 14 September 2011 due to no significant pharmacological effects (safety/PD/efficacy) through 25 mg/kg cohort, the T1/2 based on VEGF binding was shorter than expected and the current and/or higher doses were not considered feasible for further development. There were no safety concerns associated with the decision to terminate the program/study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed solid tumors unresponsive to current therapy or for which there is no standard therapy.
* Stage 2 only: Histologically or cytologically documented EOC or PPC with < or equal to 3 previous anti-cancer therapies, but at least 1 prior platinum containing regimen.
* Adequate coagulation, liver, and renal function.
* Candidate for Dynamic Contrast-Enhanced Magnetic Resonance Imaging [DCE-MRI] evaluation
* Eastern Cooperative Oncology Group [ECOG] performance status of 0 or 1

Exclusion Criteria:

* History of clinically significant toxicity to Vascular Endothelial Growth Factor [VEGF] inhibition.
* Evidence of bleeding problems.
* Uncontrolled hypertension.
* Patients with primary brain cancer and/or non-small cell lung cancer of squamous cell histology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Premiere Oncology of Arizona, Scottsdale, Arizona
  - Premiere Oncology, A Medical Corporation, Santa Monica, California
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1561001&StudyName=A%20Safety%2C%20Tolerability%2C%20And%20Pharmacokinetic%20Trial%20With%20CVX-241%20In%20Patients%20With%20Advanced%20Solid%20Tumors

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was planned to be conducted in 2 stages, however, no participant could reach out to Stage 2 due to discontinuations of all the participants in Stage 1.
Groups:
- CVX-241 (PF-05057459) 0.3 mg/kg: CVX-241 (PF-05057459) 0.3 mg/kg (milligram per kilogram) intravenous (IV) infusions once-weekly in 4 week cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons.
- CVX-241 (PF-05057459) 1 mg/kg: CVX-241 (PF-05057459) 1 mg/kg intravenous (IV) infusions once-weekly in 4 week cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons.
- CVX-241 (PF-05057459) 3 mg/kg: CVX-241 (PF-05057459) 3 mg/kg intravenous (IV) infusions once-weekly in 4 week cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons.
- CVX-241 (PF-05057459) 6 mg/kg: CVX-241 (PF-05057459) 6 mg/kg intravenous (IV) infusions once-weekly in 4 week cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons.
- CVX-241 (PF-05057459) 12 mg/kg: CVX-241 (PF-05057459) 12 mg/kg intravenous (IV) infusions once-weekly in 4 week cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons.
- CVX-241 (PF-05057459) 15 mg/kg: CVX-241 (PF-05057459) 15 mg/kg intravenous (IV) infusions once-weekly in 4 week cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons.
- CVX-241 (PF-05057459) 18 mg/kg: CVX-241 (PF-05057459) 18 mg/kg intravenous (IV) infusions once-weekly in 4 week cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons.
- CVX-241 (PF-05057459) 25 mg/kg: CVX-241 (PF-05057459) 25 mg/kg intravenous (IV) infusions once-weekly in 4 week cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons.
Period: Overall Study
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Started | 3 | 3 | 4 | 4 | 4 | 4 | 4 | 5
Treated | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 4 | 4 | 4 | 4 | 5
Not completed — Objective progression or relapse | 3 | 3 | 0 | 1 | 2 | 2 | 1 | 4
Not completed — Global deterioration of health status | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — No longer willing to continue | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all randomized subjects who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 5 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (8.54) | 55.0 (11.27) | 64.7 (2.52) | 58.8 (6.90) | 66.0 (9.13) | 55.5 (10.66) | 58.0 (7.75) | 60.6 (10.60) | 60.4 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 3 | 2 | 2 | 3 | 2 | 17
  Male | 1 | 1 | 2 | 1 | 2 | 2 | 1 | 3 | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD was defined as highest dose level for which no more than 1 participant in a dose cohort experienced dose limiting toxicity (DLT). DLT was defined as any of the following events occurring during the first 28 days of study medication and considered at least possibly-related to study medication: any grade 3 or 4 clinically-relevant non-hematologic toxicity, any clinically-significant grade 2 non-hematologic toxicity that requires 14 days to resolve (to grade 1).
Time Frame: Stage 1: Baseline up to Day 28 (end of cycle 1)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Due to premature termination of the study MTD could not be assessed.
Groups:
- All Participants: All participants who received CVX-241 (PF-05057459) 0.3, 3, 6, 12, 15, 18, 25 mg/kg (milligram per kilogram) intravenous (IV) infusions once-weekly in four-week cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons.
Arm/Group | All Participants
Number analyzed (Participants) | 0

2. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Description: RP2D was the highest dose where 0 of 3 or less than (<2) out of 6 participants experience a DLT. DLT was defined as any of the following events occurring during the first 28 days of study medication and considered at least possibly-related to study medication: any grade 3 or 4 clinically-relevant non-hematologic toxicity, any clinically-significant grade 2 non-hematologic toxicity that requires 14 days to resolve (to grade 1).
Time Frame: Stage 1: Baseline up to Day 28 (end of cycle 1)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Due to premature termination of the study RP2D could not be assessed.
Groups:
- All Participants: All participants who received CVX-241 (PF-05057459) 0.3, 3, 6, 12, 15, 18, 25 mg/kg intravenous (IV) infusions once-weekly in 4 week cycles until disease progression, unacceptable toxicity, or withdrawal for other reasons.
Arm/Group | All Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT was defined as any of the following events occurring during the first 28 days of study medication and considered at least possibly-related to study medication: any grade 3 or 4 clinically-relevant non-hematologic toxicity, any clinically-significant grade 2 non-hematologic toxicity that requires 14 days to resolve (to grade 1).
Time Frame: Stage 1: Baseline up to Week 4
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 5
participants | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0

4. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) or Serious Adverse Events (SAEs)
Description: Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. AEs included SAEs and non-SAEs that occurred during the study.
Time Frame: Baseline up to 28 days after last dose of study medication (last dose = up to Cycle 39)
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Data for Stage 2 is not reported due to early termination of the study.
Measure: Number; unit: participants
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 5
participants
  TEAE | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 5
  SAE | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2

5. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUCinf]
Description: AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞)u for unbound drug. It is obtained from AUC (0 - t)u plus AUC (t - ∞)u for unbound drug. Study drug was analysed using serum Angiopoietin-2 (Ang2) and plasma Vascular Endothelial Growth Factor (VEGF).
Time Frame: Pre-dose, 1, 2, 4, 6 hours post dose at Day 1 of cycle 1
Population: Safety analysis set included all randomized participants who received at least 1 dose of study medication. Here "n" signifies those participants who were evaluable for this measure at specified time points for each arm, respectively. Data for Stage 2 is not reported due to early termination of the study.
Measure: Geometric Mean (Standard Deviation); unit: nanogram*hours per milliliter (ng*hr/mL)
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 5
nanogram*hours per milliliter (ng*hr/mL)
  VEGF Binding: Cycle1/Day 1 (n=3,3,3,4,4,3,4,5) | 343000 (113710) | 1369000 (285830) | 3719000 (477910) | 10720000 (1598800) | 16330000 (4423000) | 26510000 (4011200) | 14550000 (3040800) | 29690000 (12366000)
  Ang2 Binding: Cycle1/Day 1 (n=3,1,1,3,3,1,2,2) | 582900 (609300) | NA (NA) — Data was not reported, since the same was not collected if participants were less than (<) 3, as planned. | NA (NA) — Data was not reported, since the same was not collected if participants were <3, as planned. | 12850000 (4116800) | 21720000 (5152000) | NA (NA) — Data was not reported, since the same was not collected if participants were <3 as planned. | NA (NA) — Data was not reported, since the same was not collected if participants were <3, as planned. | NA (NA) — Data was not reported, since the same was not collected if participants were <3, as planned.

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Study drug was analysed using serum Angiopoietin-2 (Ang2) and plasma Vascular Endothelial Growth Factor (VEGF).
Time Frame: Pre-dose, 1, 2, 4, 6 hours post dose at Day 1, Day 22 of cycle 1
Population: Safety analysis set included all randomized participants who received at least one dose of study medication. Here "n" signifies those participants who were evaluable for this measure at specified time points for each arm, respectively. Data for Stage 2 is not reported due to early termination of the study.
Measure: Geometric Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 5
nanogram per milliliter (ng/mL)
  VEGF Binding: Cycle1/Day 1 (n=3,3,3,4,4,4,4,5) | 6666 (1118.6) | 27160 (5159.8) | 60740 (3404.4) | 201400 (34298) | 306700 (49936) | 401700 (69776) | 247900 (39013) | 464400 (82330)
  VEGF Binding: Cycle1/Day 22 (n=3,3,3,3,4,4,4,5) | 7526 (1382.5) | 37210 (12217) | 64610 (6128.6) | 225200 (53613) | 350500 (53370) | 489800 (197080) | 304200 (39449) | 567300 (133310)
  Ang2 Binding: Cycle1/Day 1 (n=3,3,3,4,4,4,4,5) | 8056 (1944.3) | 35490 (14492) | 69320 (17218) | 180800 (34121) | 313400 (52077) | 455900 (89920) | 277800 (26998) | 459100 (103170)
  Ang2 Binding: Cycle1/Day 22 (n=3,3,3,3,4,4,4,5) | 9454 (2011.0) | 50840 (14031) | 81410 (4650.8) | 256000 (83540) | 404400 (60272) | 607500 (139340) | 406800 (60690) | 600200 (183030)

7. Secondary Outcome: Minimum Observed Plasma Trough Concentration (Cmin)
Time Frame: Pre-dose, 1, 2, 4, 6 hours post dose at Day 1, Day 22 of cycle 1
Population: Due to premature termination of the study Cmin data were not calculated, only certain pre-specified exposure related non compartmental pharmacokinetics (PK) parameters were calculated.
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Systemic Clearance (CL)
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. Due to premature termination of the study, only certain exposure-related noncompartmental PK parameters were calculated.
Time Frame: Pre-dose, 1, 2, 4, 6 hours post dose at Day 1, Day 22 of cycle 1
Population: Due to premature termination of the study, CL data were not calculated, only certain pre-specified exposure related non compartmental pharmacokinetics (PK) parameters were calculated.
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Plasma Decay Half-Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half. Study drug was analysed using serum Angiopoietin-2 (Ang2) and plasma Vascular Endothelial Growth Factor (VEGF).
Time Frame: Pre-dose, 1, 2, 4, 6 hours post dose at Day 1 of cycle 1
Population: Safety analysis set included all randomized participants who received at least one dose of study medication. Data for Stage 2 is not reported due to early termination of the study.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 5
hours
  VEGF Binding: Cycle1/Day 1 (n=3,3,3,4,4,3,4,5) | 44.87 (5.5411) | 47.20 (6.8986) | 50.53 (4.6544) | 45.38 (11.857) | 49.33 (6.9921) | 61.87 (8.1978) | 52.80 (8.5210) | 50.76 (10.308)
  Ang2 Binding: Cycle1/Day 1 (n=3,1,1,3,3,1,2,2) | 58.87 (8.4583) | NA (NA) — Data was not reported, since the same was not collected if participants were <3, as planned. | NA (NA) — Data was not reported, since the same was not collected if participants were <3, as planned. | 57.10 (11.898) | 62.53 (7.5871) | NA (NA) — Data was not reported, since the same was not collected if participants were <3. as planned. | NA (NA) — Data was not reported, since the same was not collected if participants were <3, as planned. | NA (NA) — Data was not reported, since the same was not collected if participants were <3, as planned.

10. Secondary Outcome: Change From Baseline in Plasma Vascular Endothelial Growth Factor (VEGF) Concentrations
Description: VEGF family consists of five glycoproteins known as VEGF-A, -B, -C, and -D, and placental growth factor (PlGF), which bind to three structurally similar receptor tyrosine kinases VEGFR1, VEGFR2, and VEGFR3. The different ligands have distinctive binding specificities for each of the receptors. In response to ligand binding, the VEGFRs activate distinct downstream signalling pathways. VEGFR2 is expressed in the vasculature and is the key mediator of VEGF-induced angiogenesis.
Time Frame: Cycle 1/Day 1, Cycle 1/Day 5, Cycle 1/Day 8, Cycle 1/Day 15, Cycle 1/Day 22, Cycle 2/Day 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 5
picogram/milliliter (pg/mL)
  CYCLE1/DAY1 (n=3,3,3,4,4,4,4,5) | 208.3 (182.51) | 731.3 (1119.40) | 308.7 (238.30) | 0.0 (0.00) | 1191.8 (1309.13) | 35.3 (70.50) | 1640.0 (1232.21) | 3596.6 (6740.70)
  CYCLE1/DAY5 (n=3,3,3,4,4,4,4,5) | 193.3 (193.00) | 826.7 (911.89) | 525.3 (282.46) | 617.3 (311.94) | 2410.3 (2133.08) | 637.5 (91.29) | 5758.8 (8595.09) | 3463.8 (5076.53)
  CYCLE1/DAY8 (n=3,3,3,4,4,4,4,5) | 255.0 (289.70) | 712.3 (752.83) | 392.3 (227.87) | 316.8 (228.54) | 2021.0 (1153.51) | 456.3 (160.88) | 4120.5 (6036.92) | 3124.4 (4529.62)
  CYCLE1/DAY15 (n=3,3,3,4,4,4,4,5) | 212.0 (367.19) | 564.7 (680.62) | 416.7 (179.06) | 432.5 (132.14) | 2426.5 (1615.67) | 434.3 (212.43) | 2416.8 (2247.30) | 2838.6 (4036.03)
  CYCLE1/DAY22 (n=3,3,3,3,4,4,4,5) | 327.7 (446.32) | 441.0 (596.73) | 544.3 (269.10) | 196.3 (73.38) | 2601.5 (1405.06) | 444.8 (231.80) | 2888.0 (3733.88) | 2447.2 (3163.16)
  CYCLE2/DAY1 (n=2,3,3,3,4,4,3,4) | 394.0 (557.20) | 414.7 (516.34) | 636.3 (298.84) | 230.0 (199.68) | 2402.5 (1582.10) | 553.3 (573.44) | 1283.0 (697.74) | 2167.8 (2947.41)

11. Secondary Outcome: Change From Baseline in Serum Angiopoietin-2 (Ang2) Concentrations
Description: Angiopoietin-2 (Ang2) and a related protein, angiopoietin-1 (Ang1) are ligands of the endothelial cell receptor Tie-2, a receptor tyrosine kinase, and are known to mediate the angiogenesis process together with VEGF and other angiogenic regulators. Ang1 stimulates the phosporylation of Tie-2, recruits pericytes to newly formed blood vessels, and promotes their maturation. Ang2 competes with Ang1 for binding of Tie-2, promotes the dissociation of pericytes, and results in unstable blood vessels. In the presence of VEGF and other angiogenic factors, endothelial cells in these unstable vessels proliferate and migrate to form new blood vessels.
Time Frame: Cycle 1/Day 1, Cycle 1/Day 5, Cycle 1/Day 8, Cycle 1/Day 15, Cycle 1/Day 22, Cycle 2/Day 1
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 5
pg/mL
  CYCLE1/DAY1 (n=3,3,3,4,4,4,4,5) | 3913.3 (701.59) | 2793.3 (1570.01) | 5756.7 (4274.81) | 3225.0 (1299.55) | 3855.0 (1749.79) | 2360.0 (477.56) | 11717.5 (15706.56) | 4570.0 (2546.22)
  CYCLE1/DAY5 (n=3,3,3,4,4,4,4,5) | 45266.7 (14202.93) | 128400 (81005.43) | 214000 (25632.01) | 272750 (97250.11) | 199750 (58025.14) | 140750 (15261.61) | 1040250 (1458899.67) | 319760 (161304.33)
  CYCLE1/DAY8 (n=3,3,3,4,4,4,4,5) | 32833.3 (14908.16) | 84933.3 (53814.16) | 195667 (39703.06) | 228000 (87089.99) | 174750 (42129.76) | 122850 (26305.07) | 788750 (1308363.19) | 332360 (175180.04)
  CYCLE1/DAY15 (n=3,3,3,3,4,4,4,5) | 32633.3 (16323.70) | 126900 (90126.63) | 195333 (54151.02) | 289333 (60302.02) | 193500 (50836.34) | 123725 (74040.32) | 754750 (1197391.99) | 208440 (148597.92)
  CYCLE1/DAY22 (n=3,3,3,3,4,4,4,5) | 36866.7 (18504.14) | 128900 (85837.11) | 262000 (67638.75) | 296000 (118000.00) | 255750 (139588.38) | 123025 (60535.41) | 786750 (1112399.32) | 223200 (150193.87)
  CYCLE2/DAY1 (n=2,3,3,3,4,4,3,4) | 46800.0 (141.42) | 130100 (90157.25) | 298000 (145578.16) | 256333 (107802.29) | 224750 (69935.09) | 132125 (75906.05) | 264000 (124755.76) | 233575 (169090.48)

12. Secondary Outcome: Number of Anti Drug Antibody Samples With Positive Anti-CVX-241 Antibodies
Description: Results were summarized for overall study population as per planned analysis.
Time Frame: Day 1 pre-dose of each cycle up to last dose of study medication (last dose = up to Cycle 39)
Population: as for outcome 9
Measure: Number; unit: samples
Arm/Group | All Participants
Number analyzed (Participants) | 30
samples | 66

13. Secondary Outcome: Objective Response Rate - Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based assessment of complete response (CR) or partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1). CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis <10 mm). No new lesions. PR was defined as >=30% decrease under baseline of the sum of diameters of all target lesions. The short aixs was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions. Stable disease was defined as not qualifying for CR, PR, and Progressive Disease.
Time Frame: Every 8 weeks from start of treatment until last dose of study medication (last dose = up to Cycle 39)
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 5
percentage of participants
  Complete Response (CR) | 0 (701.59) | 0 (1570.01) | 0 (4274.81) | 0 (1299.55) | 0 (1749.79) | 0 (477.56) | 0 (15706.56) | 0 (2546.22)
  Partial Response (PR) | 0 (14202.93) | 0 (81005.43) | 0 (25632.01) | 0 (97250.11) | 0 (58025.14) | 25.0 (15261.61) | 0 (1458899.67) | 0 (161304.33)

14. Secondary Outcome: Participants WithTumor Response of CA-125 Epithelial Ovarian Cancer (EOC)/ Primary Peritoneal Cancer (PPC)
Description: Participants with epithelial ovarian cancer or primary peritoneal cancer having CA-125 levels greater than 2x the upper limit of normal, 2 weeks prior to starting therapy were evaluated for CA-125 response and response is defined as a 50% decrease in CA-125 from a pre-treatment sample. The response was confirmed and maintained for at least 28 days. CA-125 response was calculated as intervening samples and the 28-day confirmatory sample must be less than or equal to (within assay variability of 10%) the previous sample Progression or recurrence based on serum CA-125 is defined according to the participants baseline levels.
Time Frame: Stage 2 every cycle
Population: Results are not reported for this measure, as, none of the participants could reach out to Stage 2 due to discontinuations of all the participants in Stage 1.
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Participants With Reduction in Tumor Vascular Permeability: Blood Flow and Blood Volume as Measured by Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI)
Description: DCE-MRI is a non-invasive method that provides a functional assessment of microvasculature. The technique can measure changes in vascular permeability, extracellular, and extravascular and vascular volumes. Based on its ability to detect vascular changes, DCE-MRI has recently been evaluated as a biomarker of drug efficacy in clinical trials of angiogenesis inhibitors. Assessment of DCE-MRI started at the 3.0 mg/kg dose cohort.
Time Frame: Stage 2 predose up to end of study
Population: as for outcome 14
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as non-serious in another subject, or one subject may have experienced both a serious and non-serious event during the study.
Arm/Group | CVX-241 (PF-05057459) 0.3 mg/kg | CVX-241 (PF-05057459) 1 mg/kg | CVX-241 (PF-05057459) 3 mg/kg | CVX-241 (PF-05057459) 6 mg/kg | CVX-241 (PF-05057459) 12 mg/kg | CVX-241 (PF-05057459) 15 mg/kg | CVX-241 (PF-05057459) 18 mg/kg | CVX-241 (PF-05057459) 25 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 2/4 | 0/4 | 1/4 | 1/4 | 2/5
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 4/4 | 4/4 | 4/4 | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVX-241 (PF-05057459) 0.3 mg/kg (N=3) | CVX-241 (PF-05057459) 1 mg/kg (N=3) | CVX-241 (PF-05057459) 3 mg/kg (N=3) | CVX-241 (PF-05057459) 6 mg/kg (N=4) | CVX-241 (PF-05057459) 12 mg/kg (N=4) | CVX-241 (PF-05057459) 15 mg/kg (N=4) | CVX-241 (PF-05057459) 18 mg/kg (N=4) | CVX-241 (PF-05057459) 25 mg/kg (N=5)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Drug withdrawal syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CVX-241 (PF-05057459) 0.3 mg/kg (N=3) | CVX-241 (PF-05057459) 1 mg/kg (N=3) | CVX-241 (PF-05057459) 3 mg/kg (N=3) | CVX-241 (PF-05057459) 6 mg/kg (N=4) | CVX-241 (PF-05057459) 12 mg/kg (N=4) | CVX-241 (PF-05057459) 15 mg/kg (N=4) | CVX-241 (PF-05057459) 18 mg/kg (N=4) | CVX-241 (PF-05057459) 25 mg/kg (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal rigidity (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Early satiety (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 2 | 0 | 1 | 1 | 2 | 2 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0 | 2 | 1 | 1 | 2 | 2
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Breast discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Capillaritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 2

LIMITATIONS AND CAVEATS:
The study was terminated early by the sponsor due to lack of significant pharmacological effects (safety/Pharmacodynamics/efficacy) through 25 mg/kg cohort. Hence, no participant could reach out to Stage 2.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.